CLINICAL TRIAL: NCT05590793
Title: A Multicentre, Open-label, Single-arm Study to Investigate the Efficacy and Safety of Triptorelin Pamoate 22.5 mg 6-month Formulation in Chinese Patients With Locally Advanced or Metastatic Prostate Cancer
Brief Title: Effects of Triptorelin Pamoate 6-month When Given to Adult Chinese Participants With Advanced Cancer in the Prostate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-CN-52014-237; CTR20221796 (Registry Identifier: ChinaDrugTrial.org)
Record Dates: First submitted 2022-10-14; First posted 2022-10-21 (Actual); Results first posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Advanced Prostate Cancer; Metastatic Prostate Cancer; Locally Advanced Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Triptorelin Pamoate; Salts

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Triptorelin pamoate 22.5 mg 6-month formulation (Experimental): All enrolled participants will receive one intramuscular (i.m.) injection of containing 22.5 mg 6-month formulation triptorelin pamoate on Day 1.
  Interventions: Drug: Triptorelin pamoate (embonate) salt

INTERVENTIONS:
Drug: Triptorelin pamoate (embonate) salt — Triptorelin pamoate 22.5 mg (6-month formulation), i.m. injection, single dose on Day 1.
  Other Names: Dipherelin

SUMMARY:
The main aim of this study is to assess the effectiveness and safety of the 6-month formulation of triptorelin pamoate in Chinese participants with locally advanced or metastatic cancer of the prostate. Participants will receive 1 injection of triptorelin pamoate 6-month formulation.

ELIGIBILITY:
Inclusion Criteria :

* Participant is capable of giving signed informed consent
* Participant must be over 18 years of age, at the time of signing the informed consent.
* Has a histologically or cytologically confirmed adenocarcinoma, locally advanced or metastatic prostate cancer. Or participant has PSA recurrence after curative treatment and be a candidate for androgen deprivation therapy (ADT).
* Has serum testosterone level >150 ng/dL (> 5.2 nmol/L).
* Has expected survival time ≥12 months according to the investigator's assessment.
* Has Eastern Cooperative Oncology Group (ECOG) performance status score ≤1

Exclusion Criteria :

* Risk of a serious complication in the case of tumour flare
* Presence of another neoplastic lesion or brain metastases.
* Previous history of QT prolongation or concomitant use of medicinal products known to prolong the QT interval or with a known risk of torsades de pointes.
* Metastatic hormone-sensitive prostate cancer with high tumour burden.
* Metastatic castration-resistant prostate cancer.
* Previous surgical castration.
* Previous hormone therapy (including abiraterone) for prostate cancer within 6 months prior to study start.
* Previous cytotoxic chemotherapy treatment within 6 months prior to study screening.
* Use of finasteride or dutasteride within 2 months prior to study screening.
* Previous hypophysectomy or adrenalectomy
* Any current use or use within 6 months prior to treatment start of medications which are known to affect the metabolism and/or secretion of androgenic hormones: ketoconazole, aminoglutethimide, oestrogens and antiandrogens.
* Current use of systemic or inhaled corticosteroids (topical application permitted).
* Any previous use of traditional Chinese medicine or herbal products within 1 month prior to study screening or planned use during the study of products, which are known to have cytotoxic effect or affect the metabolism and/or secretion of androgenic hormones
* Participation in another study with an investigational drug or treatment within 3 months prior to study screening or within 5 drug half-lives of the investigational drug (whichever is the longer).
* Severe kidney or liver impairment (creatinine >2 x upper limit of normal (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) >3 x ULN).
* Any concomitant disorder or resulting therapy that is likely to interfere with participant compliance, the i.m. administration of the drug or with the study in the opinion of the investigator.
* Known hypersensitivity to triptorelin or any of its excipients, GnRH, other GnRH agonist/analogues.
* Known active use of recreational drug or alcohol dependence in the opinion of the investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only Male is enrolled
Enrollment: 195 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical, Director, Study Director — Ipsen
Locations (36):
- China (36):
  - Affiliated Hospital of Hebei University, Baoding
  - Beijing Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - Hunan Cancer Hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Deyang People's Hospital, Deyang
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Qilu Hospital of Shandong University, Jinan
  - Shandong Provincial Hospital, Jinan
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Ningbo First Hospital, Ningbo
  - Fudan University Shang Hai Cancer Center, Shanghai
  - Shanghai Fifth People's Hospital, Shanghai
  - Shanghai Tongji Hospital, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The First Hospital of China Medical University, Shenyang
  - Peking University Shenzhen Hospital, Shenzhen
  - Suining Central Hospital, Suining
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin Cancer Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The First Affiliated Hospital of Wannan Medical College, Wuhu
  - The Second Affiliated Hospital of Wannan Medical College, Wuhu
  - Wuxi People's Hospital, Wuxi
  - Northern Jiangsu People's Hospital, Yangzhou
  - Subei People's Hospital, Yangzhou
  - Yantai Yuhuangding Hospital, Yantai
  - Henan Cancer Hospital, Zhengzhou
  - Zigong First People's Hospital, Zigong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
  Any requests should be submitted to www.vivli.org for assessment by an independent scientific review board.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and EU or after the primary manuscript describing the results has been accepted for publication, whichever is later.
Access Criteria: Further details on Ipsen's sharing criteria, eligible studies and process for sharing are available here (https://vivli.org/members/ourmembers/).
URL: https://vivli.org/members/ourmembers

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase IIIb, open-label, single arm study was conducted at 27 investigational sites in participants with locally advanced or metastatic prostate cancer.
Pre-assignment Details: The study consisted of a 4-week screening period, single dose study intervention administration on Day 1 and an end of study on Day 169. A subset of participants had a more extensive sampling during the study to evaluate pharmacokinetics (PK) and pharmacodynamics (PD). A total of 195 participants were enrolled in the study.
Groups:
- Triptorelin Pamoate: Participants received a single dose of triptorelin pamoate 22.5 milligrams (mg) intramuscular (IM) injection on Day 1.
Period: Overall Study
Arm/Group | Triptorelin Pamoate
Started | 195
Completed | 188
Not Completed | 7
Not completed — Withdrawal by Subject | 6
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who received the single dose of study intervention.
Groups:
- Triptorelin Pamoate: Participants received a single dose of triptorelin pamoate 22.5 mg IM injection on Day 1.
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 195
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 195

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Castrate Levels of Serum Testosterone on Day 29
Description: Blood samples were collected to determine the serum testosterone concentrations using a validated, specific and sensitive liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Achievement of testosterone castration was defined as serum testosterone level <50 nanograms per deciliter (ng/dL) or 1.735 nanomoles/liter (nmol/L). Percentages are rounded off to the tenth decimal place.
Time Frame: Day 29
Population: The full analysis set (FAS) included all treated participants who completed the study or were a treatment failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 188
percentage of participants | 99.5 [97.1 to 100.0]

2. Primary Outcome: Percentage of Participants Who Maintained the Castrate Levels From Week 8 to Week 24
Description: Blood samples were collected to determine the serum testosterone concentrations using a validated, specific and sensitive LC-MS/MS method. Maintenance of castration was defined as serum testosterone level <50 ng/dL or 1.735 nmol/L.
Time Frame: From Week 8 to Week 24
Population: The FAS included all treated participants who completed the study or were a treatment failure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 188
percentage of participants | 100 [98.1 to 100.0]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (TESAEs) and Treatment-Emergent Adverse Events of Local Tolerance
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An SAE was any untoward medical occurrence that, at any dose, resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital abnormality/birth defect, or any other medically important event. TEAEs were AEs with start date on or after the date of study intervention administration and up to 24 weeks after date of first dose of treatment. Local tolerance was assessed 2 hours (+/-15 minutes) after the single injection of 6-month formulation triptorelin by examination of injection site for signs including but not limited to tenderness, erythema, swelling, hematoma, rash, pain, itching and induration.
Time Frame: From the first dose of study intervention (Day 1) up to end of study visit (Week 24), approximately 169 days
Population: The safety set included all participants who received the single dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 195
Participants
  Any TEAEs | 160
  Any TESAEs | 8
  TEAEs of Local Tolerance | 7

4. Secondary Outcome: Percent Change From Baseline in Prostate Specific Antigen (PSA) at Weeks 12 and 24
Description: Blood samples were collected for the measurement of plasma PSA concentrations. Percent change in PSA was defined as the absolute value of difference between the PSA values at Week 12 and Week 24 and the baseline value divided by the baseline value. Baseline was defined as the last non-missing measurement taken prior to first study intervention administration.
Time Frame: Baseline (Day 1), Weeks 12 and 24
Population: The FAS included all treated participants who completed the study or were a treatment failure. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 187
percent change
  Week 12 | -90.6815 (10.8057)
  Week 24: number analyzed (Participants) | 186
  Week 24 | -92.1673 (12.2853)

5. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of Triptorelin Pamoate
Description: Blood samples were collected at specified timepoints for the assessment of tmax of triptorelin pamoate. The PK parameters were performed using non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96 and 168 hours post-dose on Day 1, Days 15, 22, 29, 57, 85, 113, 141 and 169
Population: The rich PK analysis set included all participants in the rich PK/PD subset who received 1 dose of study intervention, had no major protocol deviations affecting the PK variables, and who had a sufficient number of plasma concentrations to estimate the main PK parameters (maximum observed plasma drug concentration [Cmax], tmax and area under the plasma concentration time curve [AUC]).
Measure: Median (Full Range); unit: hour
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 12
hour | 2.95 [1.93 to 11.5]

6. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Triptorelin Pamoate
Description: Blood samples were collected at specified timepoints for the assessment of Cmax of triptorelin pamoate. The PK parameters were performed using non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96 and 168 hours post-dose on Day 1, Days 15, 22, 29, 57, 85, 113, 141 and 169
Population: The rich PK analysis set included all participants in the rich PK/PD subset who received 1 dose of study intervention, had no major protocol deviations affecting the PK variables, and who had a sufficient number of plasma concentrations to estimate the main PK parameters (Cmax, tmax and AUC).
Measure: Mean (Standard Deviation); unit: ng/milliliter (mL)
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 12
ng/milliliter (mL) | 44.5 (17.5)

7. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to the Visit on Day 169 (AUC0-169) of Triptorelin Pamoate
Description: Blood samples were collected at specified timepoints for the assessment of AUC0-169 of triptorelin pamoate. The PK parameters were performed using non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96 and 168 hours post-dose on Day 1, Days 15, 22, 29, 57, 85, 113, 141 and 169
Population: The rich PK analysis set included all participants in the rich PK/PD subset who received 1 dose of study intervention, had no major protocol deviations affecting the PK variables, and who had a sufficient number of plasma concentrations to estimate the main PK parameters (Cmax, tmax and AUC). Only those participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 9
ng*day/mL | 51.7 (22.9)

8. Secondary Outcome: Area Under the Plasma Concentration Time Curve From Time 0 to the Last Quantifiable Concentration (AUClast) of Triptorelin Pamoate
Description: Blood samples were collected at specified timepoints for the assessment of AUClast of triptorelin pamoate. The PK parameters were performed using non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 3, 4, 6, 8, 12, 24, 48, 96 and 168 hours post-dose on Day 1, Days 15, 22, 29, 57, 85, 113, 141 and 169
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: ng*day/mL
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 12
ng*day/mL | 46.3 (22.1)

9. Secondary Outcome: Time to Maximum Observed Plasma Concentration of Testosterone
Description: Blood samples were collected at specified timepoints for the assessment of tmax of testosterone. The PD parameters were performed using non-compartmental analysis.
Time Frame: Pre-dose on Day 1 and Days 2, 3, 5, 8, 15, 22, 29, 57, 85, 113, 141 and 169
Population: The rich PD analysis set included all participants in the rich PK/PD subset who had a sufficient number of PD (testosterone) measurements to estimate the main PD parameters (Cmax, tmax and time to castration [tcast]).
Measure: Median (Full Range); unit: day
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 12
day | 2.00 [0 to 4.02]

10. Secondary Outcome: Maximum Observed Plasma Concentration of Testosterone
Description: Blood samples were collected at specified timepoints for the assessment of Cmax of testosterone. The PD parameters were performed using non-compartmental analysis.
Time Frame: Pre-dose on Day 1 and Days 2, 3, 5, 8, 15, 22, 29, 57, 85, 113, 141 and 169
Population: The rich PD analysis set included all participants in the rich PK/PD subset who had a sufficient number of PD (testosterone) measurements to estimate the main PD parameters (Cmax, tmax and tcast).
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 12
nmol/L | 21.9 (6.55)

11. Secondary Outcome: Time to Castration of Testosterone
Description: Blood samples were collected at specified timepoints for the assessment of tcast of testosterone. tcast was defined as time to reach serum testosterone level <50 ng/dL or 1.735 nmol/L. The PD parameters were performed using non-compartmental analysis.
Time Frame: Pre-dose on Day 1 and Days 2, 3, 5, 8, 15, 22, 29, 57, 85, 113, 141 and 169
Population: as for outcome 10
Measure: Median (Full Range); unit: day
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 12
day | 19.3 [14.5 to 25.3]

12. Secondary Outcome: Plasma Concentrations of Triptorelin Pamoate
Description: Blood samples were collected at specified timepoints for the assessment of plasma concentration of triptorelin pamoate.
Time Frame: Pre-dose on Day 1 and post-dose at Weeks 4, 8, 12, 16, 20 and 24
Population: The population PK analysis set included all participants who received 1 dose of triptorelin and who had at least 1 triptorelin plasma concentration and no major protocol deviations affecting PK variables. Only participants with data collected at specified timepoints are reported.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 190
ng/mL
  Day 1: number analyzed (Participants) | 1
  Day 1 | NA (NA) — NA indicates that data was not estimable as the values were below the lower limit of quantification (LLOQ). The LLOQ value was 0.0100 ng/mL.
  Week 4 | 0.0743 (0.0342)
  Week 8: number analyzed (Participants) | 187
  Week 8 | 0.1236 (0.0536)
  Week 12: number analyzed (Participants) | 186
  Week 12 | 0.0602 (0.0551)
  Week 16: number analyzed (Participants) | 181
  Week 16 | 0.1555 (0.0974)
  Week 20: number analyzed (Participants) | 178
  Week 20 | 0.0607 (0.0401)
  Week 24: number analyzed (Participants) | 161
  Week 24 | 0.0249 (0.0225)

13. Secondary Outcome: Serum Concentrations of Testosterone
Description: Blood samples were collected at specified timepoints for the assessment of serum concentration of testosterone.
Time Frame: Pre-dose on Day 1 and post-dose at Weeks 4, 8, 12, 16, 20 and 24
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Triptorelin Pamoate
Number analyzed (Participants) | 188
nmol/L
  Day 1 | 17.0506 (7.0323)
  Week 4 | 0.5602 (0.2749)
  Week 8: number analyzed (Participants) | 187
  Week 8 | 0.3294 (0.1513)
  Week 12: number analyzed (Participants) | 187
  Week 12 | 0.3281 (0.1416)
  Week 16: number analyzed (Participants) | 186
  Week 16 | 0.3334 (0.1539)
  Week 20: number analyzed (Participants) | 184
  Week 20 | 0.3404 (0.1580)
  Week 24 | 0.3828 (0.1899)

ADVERSE EVENTS:
Time Frame: TEAEs are reported from the first dose of study intervention (Day 1) up to end of study visit (Week 24), approximately 169 days
Description: The safety set included all participants who received the single dose of study intervention.
Arm/Group | Triptorelin Pamoate
All-Cause Mortality (participants affected / at risk) | 0/195
Serious Adverse Events (participants affected / at risk) | 8/195
Other Adverse Events (participants affected / at risk) | 90/195
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate (N=195)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Lacunar infarction (Nervous system disorders) | 1 (1)
Skin oedema (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triptorelin Pamoate (N=195)
Anaemia (Blood and lymphatic system disorders) | 16 (16)
Pyrexia (General disorders) | 11 (13)
Upper respiratory tract infection (Infections and infestations) | 18 (25)
Nasopharyngitis (Infections and infestations) | 15 (19)
Alanine aminotransferase increased (Investigations) | 12 (14)
Aspartate aminotransferase increased (Investigations) | 10 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (26)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 15 (32)
Hot flush (Vascular disorders) | 11 (11)
Hypertension (Vascular disorders) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT05590793/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-24): https://cdn.clinicaltrials.gov/large-docs/93/NCT05590793/SAP_001.pdf